CLINICAL TRIAL: NCT07198542
Title: Treatment of Somatic Symptom Disorder With Transcutaneous Cervical Vagus Nerve Stimulation and Transcutaneous Auricular Vagus Nerve Stimulation: A Crossover Randomized Controlled Trial
Brief Title: Treatment of SSD With tcVNS and taVNS
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Industrial Technology Research Institute, Taiwan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 202411116DIND
Record Dates: First submitted 2025-09-21; First posted 2025-09-30 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Somatic Symptom Disorder; Anxiety; Depression; Transcutaneous Vagus Nerve Stimulation; Neuromodulation
Keywords: Somatic Symptom Disorder; Transcutaneous Vagus Nerve Stimulation; Neuromodulation; Anxiety; Depression
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: This is a single-blind study. In addition to the Outcomes Assessor, the Statistical Analyst will also be blinded to the treatment allocation. The analyst will receive a dataset with treatment groups coded (e.g., 'Group A', 'Group B') and will perform the statistical analysis without knowledge of which group corresponds to which intervention. The allocation code will be revealed only after the primary analysis is complete and the results have been confirmed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: gammaCore then Nurosym (Experimental): Participants assigned to this sequence will first receive active transcutaneous cervical vagus nerve stimulation (tcVNS) using the gammaCore device. This initial treatment period consists of 10 daily sessions (approx. 20 minutes each) over 2 weeks, followed by a 1-week follow-up assessment. After a 1-week washout period, participants will cross over to the second treatment period. In this period, they will receive active transcutaneous auricular vagus nerve stimulation (taVNS) using the Nurosym device for 10 daily 30-minute sessions over 2 weeks, followed by a final 1-week follow-up assessment.
  Interventions: Device: gammaCore Sapphire; Device: Nurosym
- Group B: Nurosym then gammaCore (Experimental): Participants assigned to this sequence will first receive active transcutaneous auricular vagus nerve stimulation (taVNS) using the Nurosym device. This initial treatment period consists of 10 daily 30-minute sessions over 2 weeks, followed by a 1-week follow-up assessment. After a 1-week washout period, participants will cross over to the second treatment period. In this period, they will receive active transcutaneous cervical vagus nerve stimulation (tcVNS) using the gammaCore device for 10 daily sessions (approx. 20 minutes each) over 2 weeks, followed by a final 1-week follow-up assessment.
  Interventions: Device: gammaCore Sapphire; Device: Nurosym

INTERVENTIONS:
Device: gammaCore Sapphire — This intervention utilizes transcutaneous cervical Vagus Nerve Stimulation (tcVNS). A conductive gel is applied to the device's stimulation surfaces. The device is then placed on the neck over the vagus nerve. The daily treatment protocol consists of three consecutive 2-minute stimulations on the left side of the neck, with a 30-60 second interval between each stimulation. After a brief rest of approximately one minute, the same procedure is repeated on the right side of the neck. The total daily session duration is approximately 20 minutes. Stimulation intensity is individually titrated for each participant to a level that is perceptible but not painful. This regimen is administered once daily for 10 sessions over a 2-week period.
  Other Names: Transcutaneous cervical Vagus Nerve Stimulation; tcVNS
Device: Nurosym — This intervention utilizes transcutaneous auricular Vagus Nerve Stimulation (taVNS). The device consists of an earpiece electrode that is clipped onto the left tragus. A small amount of water is applied to the skin for conductivity. The daily treatment protocol consists of one continuous 30-minute stimulation session. Stimulation intensity is individually titrated for each participant to a level that is perceptible but not painful. This regimen is administered once daily for 10 sessions over a 2-week period.
  Other Names: Transcutaneous auricular Vagus Nerve Stimulation; taVNS

SUMMARY:
This study aims to compare two non-invasive nerve stimulation devices, gammaCore and Nurosym, to find out which one is more effective in reducing physical discomfort and health-related anxiety in patients with Somatic Symptom Disorder, a condition where individuals experience significant physical symptoms and have excessive thoughts and worries about their health.

Participants in this study will receive treatment using both devices at different times. Both devices work by sending mild electrical pulses through the skin to stimulate the vagus nerve, a major nerve that helps regulate body functions. One device (gammaCore) is placed on the neck, while the other (Nurosym) is worn on the ear.

The order in which a participant receives the two treatments will be decided by chance, like flipping a coin. Each treatment period will last for two weeks, with a one-week break in between. Over the course of the study (about 8 weeks), participants will visit the hospital for treatment sessions and to complete questionnaires and have non-invasive measurements of body responses, such as heart rate variability.

DETAILED DESCRIPTION:
Official Title: Treatment of Somatic Symptom Disorder with Transcutaneous Cervical Vagus Nerve Stimulation and Transcutaneous Auricular Vagus Nerve Stimulation: A Crossover Randomized Controlled Trial.

Study Design: This is a single-center, randomized, single-blind (assessor- and analyst-blinded), crossover clinical trial designed to compare the efficacy of two transcutaneous vagus nerve stimulation (tVNS) devices in patients with Somatic Symptom Disorder (SSD). Participants will be randomly assigned to one of two sequences: (A) Nurosym followed by gammaCore, or (B) gammaCore followed by Nurosym. Each intervention phase consists of 10 daily stimulation sessions administered over a 2-week period (Monday-Friday), followed by a 1-week follow-up assessment. A 1-week washout period will separate the two intervention phases.

Primary Objectives: The primary objective is to compare the efficacy of transcutaneous cervical VNS (tcVNS) delivered by the gammaCore device versus transcutaneous auricular VNS (taVNS) delivered by the Nurosym device on the core symptoms of SSD. This will be measured by the change in scores on the Patient Health Questionnaire-15 (PHQ-15) for somatic symptom severity and the Health Anxiety Questionnaire (HAQ) for health anxiety.

Secondary Objectives: Secondary objectives include evaluating the effects of both treatments on depression, anxiety, worry, and physiological markers of autonomic nervous system function (e.g., heart rate variability, skin conductance, finger temperature). The study will also explore factors that may predict treatment response.

Interventions:

Device 1 (gammaCore): Delivers tcVNS. The device will be applied to the neck over the vagus nerve. The daily session involves three 2-minute stimulations on the left side of the neck, followed by three 2-minute stimulations on the right side, for a total daily treatment time of approximately 20 minutes.

Device 2 (Nurosym): Delivers taVNS. The device uses an earpiece placed on the left tragus to stimulate the auricular branch of the vagus nerve. The daily treatment consists of one continuous 30-minute session.

Stimulation intensity for both devices will be individually titrated for each participant to a level described as a "clear but not uncomfortable or painful sensation".

Outcome Measures:

Primary Endpoints: The primary endpoints are the change from baseline (Day 1 or Day 29) to the 1-week follow-up assessment (Day 19 or Day 47) in PHQ-15 and HAQ scores for each treatment period .

Secondary Endpoints: Secondary outcome measures include the change from baseline to all subsequent assessment points (e.g., Day 5, Day 12, Day 19) in the Beck Depression Inventory-II (BDI-II), Beck Anxiety Inventory (BAI), Penn State Worry Questionnaire (PSWQ), and various physiological parameters. Safety will be assessed by monitoring adverse events throughout the study.

ELIGIBILITY:
Inclusion Criteria:

1. Meets the diagnostic criteria for Somatic Symptom Disorder (SSD) according to the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5), as determined by a diagnostic interview with a board-certified psychiatrist.
2. The participant must be receiving stable, routine medical care throughout the trial period.
3. No adjustments to psychiatric or cardiovascular medications for at least one week prior to the start of the study.

Exclusion Criteria:

1. Age below 18 or above 65 years.
2. Presence of psychotic symptoms, such as in comorbid schizophrenia.
3. Significant cognitive impairment (e.g., diagnosed dementia or intellectual disability) or difficulty completing the study questionnaires.
4. History of cervical vagotomy.
5. Presence of severe cardiovascular diseases, including: clinically significant tachycardia (resting heart rate >100 bpm) or bradycardia (resting heart rate <60 bpm); clinically significant hypertension (systolic >160 mmHg or diastolic >100 mmHg) or hypotension (blood pressure <90/60 mmHg or mean arterial pressure <65 mmHg); severe coronary artery disease; carotid atherosclerosis or stenosis; aneurysm; congestive heart failure; severe cardiac arrhythmias (e.g., prolonged QT interval, second- or third-degree atrioventricular block, atrial fibrillation, atrial flutter, recent ventricular tachycardia or fibrillation, clinically significant premature ventricular contractions); or myocardial infarction within the last five years.
6. Presence of severe neurological conditions, including severe head trauma, history of epilepsy, brain tumor, or cerebral hemorrhage.
7. Current diagnosis of cancer.
8. Presence of any active implanted medical devices (e.g., cochlear implant, ventricular shunt, implantable vagus nerve stimulator, pacemaker) or non-active implants that may interact with the nervous system (e.g., metal stents, bone plates, screws).
9. Anatomical abnormalities in the neck.
10. Currently pregnant.
11. Wearing jewelry near the tragus that cannot be removed before using the tVNS device.
12. Severe skin disease at the stimulation sites.
13. Known allergy to conductive gel materials.
14. Any other major medical condition that, in the investigator's judgment, could potentially affect the safety or efficacy of vagus nerve stimulation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-11-17 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Somatic Symptom Severity as Measured by the Patient Health Questionnaire-15 (PHQ-15) | Change from baseline (Day 1 for the first period; Day 29 for the second period) to the 1-week post-treatment follow-up assessment (Day 19 for the first period; Day 47 for the second period).
  The PHQ-15 is a 15-item self-report scale that assesses the severity of somatic symptoms. Each item is scored from 0 ("not bothered at all") to 2 ("bothered a lot"), resulting in a total score ranging from 0 to 30. Higher scores indicate greater somatic symptom severity. The outcome is the change in the total score from the baseline of each treatment period.
Change in Health Anxiety as Measured by the Health Anxiety Questionnaire (HAQ) | Change from baseline (Day 1 for the first period; Day 29 for the second period) to the 1-week post-treatment follow-up assessment (Day 19 for the first period; Day 47 for the second period).
  The Health Anxiety Questionnaire (HAQ) is a self-report scale used to measure the severity of health-related anxiety, including worries and beliefs about health. Total scores are calculated, with higher scores indicating a greater level of health anxiety. The outcome is the change in the total score from the baseline of each treatment period.

SECONDARY OUTCOMES:
Change in Depressive Symptom Severity as Measured by the Beck Depression Inventory-II (BDI-II) | Change from baseline (Day 1 or Day 29) to each subsequent assessment point (Day 5, Day 12, Day 19 for the first period; Day 33, Day 40, Day 47 for the second period).
  The BDI-II is a 21-item self-report inventory measuring the severity of depression. The total score ranges from 0 to 63, with higher scores indicating more severe depressive symptoms. The outcome is the change in the total score from the baseline of each treatment period.
Change in Anxiety Symptom Severity as Measured by the Beck Anxiety Inventory (BAI) | Change from baseline (Day 1 or Day 29) to each subsequent assessment point (Day 5, Day 12, Day 19 for the first period; Day 33, Day 40, Day 47 for the second period).
  The BAI is a 21-item self-report inventory measuring the severity of anxiety, particularly focusing on somatic symptoms of anxiety. The total score ranges from 0 to 63, with higher scores indicating more severe anxiety. The outcome is the change in the total score from the baseline of each treatment period.
Change in General Worry as Measured by the Penn State Worry Questionnaire (PSWQ) | Change from baseline (Day 1 or Day 29) to each subsequent assessment point (Day 5, Day 12, Day 19 for the first period; Day 33, Day 40, Day 47 for the second period).
  The PSWQ is a self-report questionnaire designed to assess the trait of worry, focusing on its generality, excessiveness, and uncontrollability. Higher scores indicate a greater tendency to worry. The outcome is the change in the total score from the baseline of each treatment period.
Change in Autonomic Nervous System Function as Measured by Heart Rate Variability (HRV) | Change from baseline (Day 1 or Day 29) to each subsequent assessment point (Day 5, Day 12, Day 19 for the first period; Day 33, Day 40, Day 47 for the second period).
  HRV is a measure of the variation in time between consecutive heartbeats, used to assess cardiac autonomic regulation. Frequency-domain (e.g., High-Frequency power [HF], Low-Frequency power [LF], LF/HF ratio) and time-domain (e.g., SDNN) parameters will be analyzed.
Change in Cardiac Vagal Control as Measured by Respiratory Sinus Arrhythmia (RSA) | Change from baseline (Day 1 or Day 29) to each subsequent assessment point (Day 5, Day 12, Day 19 for the first period; Day 33, Day 40, Day 47 for the second period).
  Respiratory Sinus Arrhythmia (RSA) is the naturally occurring variation in heart rate during the breathing cycle and is considered a non-invasive index of cardiac vagal tone. It is derived from concurrently measured electrocardiogram (ECG) and respiration signals. Changes from baseline will be assessed to evaluate the intervention's effect on parasympathetic nervous system activity.
Change in Sympathetic Arousal as Measured by Skin Conductance | Change from baseline (Day 1 or Day 29) to each subsequent assessment point (Day 5, Day 12, Day 19 for the first period; Day 33, Day 40, Day 47 for the second period).
  Skin conductance measures fluctuations in the electrical characteristics of the skin, reflecting sympathetic nervous system activity. Changes from baseline will be assessed to evaluate physiological arousal.
Change in Peripheral Vasomotor Activity as Measured by Finger Temperature | Change from baseline (Day 1 or Day 29) to each subsequent assessment point (Day 5, Day 12, Day 19 for the first period; Day 33, Day 40, Day 47 for the second period).
  Peripheral skin temperature, measured at the finger, is an indicator of peripheral blood flow and is influenced by sympathetic nervous system activity. A decrease in temperature can indicate vasoconstriction associated with stress or arousal. The change from baseline will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Hao Ma, MD, Principal Investigator — Department of Psychiatry, National Taiwan University Hospital Yunlin Branch
Locations (1):
- Department of Psychiatry, National Taiwan University Hospital Yunlin Branch, Douliu, Yunlin, Taiwan

IPD SHARING:
Plan to Share IPD: No